CLINICAL TRIAL: NCT01171950
Title: CentriMag Ventricular Assist System (VAS): Treatment of Failure-to-Wean From Cardiopulmonary Bypass for Pediatric Patients
Brief Title: CentriMag Ventricular Assist System in Treating Failure-to-Wean From Cardiopulmonary Bypass for Pediatric Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PED-001
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: Thoratec Corporation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Other): All patients meeting the patient selection criteria will be treated with the CentriMag device.
  Interventions: Device: CentriMag Ventricular Assist System

INTERVENTIONS:
Device: CentriMag Ventricular Assist System — All patients will be treated with the CentriMag device for up to 30 days.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the CentriMag ventricular assist system to help pediatric patients who have experienced heart failure during surgery and cannot be removed from cardiac bypass.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 years to 16 years, inclusive
2. Inability to wean from cardiopulmonary bypass (CPB)

Exclusion Criteria:

1. Body weight < 20 kg
2. Severe aortic insufficiency
3. Unrestricted intra-cardiac communications (i.e. large VSD)
4. Pulmonary vascular resistance index (PVRI) > 10 IU
5. Presence of DIC
6. On hemodialysis (excluding hemofiltration)
7. Contraindications to systemic anticoagulation
8. Active systemic infection unresponsive to antibiotics
9. Unresolved malignancy
10. On other investigational VAS

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 30 days after device removal, or, induction of anesthesia for implant of a long-term device or heart transplant
  In patients who recover and do not go on to transplantation or a long-term device:
  • Survival 30 days after removal of the CentriMag VAS or to discharge, whichever is longer.
  In patients who do not recover:
  • Ability to be removed from the CentriMag VAS and survive to induction of anesthesia for implantation of a long-term device or heart transplantation.

SECONDARY OUTCOMES:
Evaluation of end-organ function | 30 days after device removal, or, to induction of anesthesia for implant of a long-term device or heart transplant
  Improvements in measures of end-organ function

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chatterjee, Study Director — Thoratec Corporation/Abbott